CLINICAL TRIAL: NCT00789880
Title: Analysis of the Response of Subjects With Atopic Dermatitis to Oral Vitamin D3 by Measurement of Antimicrobial Peptide Expression in Skin and Saliva
Brief Title: Analysis of Response of Subjects With Atopic Dermatitis or Psoriasis to Oral Vitamin D3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Consortium of Food Allergy Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIT ADVN CATH 03; DAIT-ADVN-CATH-03-01 Sub-study (Other: DAIT, NIAID); NCT01078259 (obsolete NCT alias)
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2013-01-22 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Atopic Dermatitis; Psoriasis
Keywords: Vitamin D3; Atopic Dermatitis; Antimicrobial Peptide Expression
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Subjects received a 21-day course of oral vitamin D3 (cholecalciferol, 4,000 international units [IU]
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Subjects received a 21-day course of oral vitamin D3-placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Administration of oral vitamin D3 at 4000IU
  Other Names: cholecalciferol
  Arms: Vitamin D3
Drug: Placebo — Administration of oral Vitamin D3 placebo
  Other Names: vitamin D3 placebo
  Arms: Placebo

SUMMARY:
This study will examine whether administration of oral Vitamin D3 given over 21 days will change the antimicrobial peptide expression in the skin or saliva of subjects with Atopic Dermatitis (AD). This study will help researchers determine if the lack of the expression of antimicrobial peptides in individuals with AD plays a role in the susceptibility to eczema vaccinatum (EV).

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is a chronic inflammatory skin disorder in which the skin becomes extremely itchy and is susceptible to recurrent skin infections. AD is thought to occur from a combination of immunological, genetic, and environmental factors. Individuals with AD are at risk for developing a severe and widely disseminated infection called eczema vaccinatum (EV). EV is caused when the live attenuated vaccinia virus in the vaccine reproduces and spreads throughout the body. Individuals with AD lack certain antimicrobial peptides, specifically cathelicidins.

This trial also includes a sub-study with individuals who have psoriasis. Psoriasis is also an immune-mediated skin disease, and is characterized by scaling skin and inflammation (pain, swelling, heat, and redness). Most psoriasis cause patches of thick, red skin with silvery scales. These patches can itch or feel sore. This sub-study will provide additional information on psoriatic responses to oral vitamin D. (Originally listed separately as ADVN-CATH-03-01).

ELIGIBILITY:
Inclusion Criteria (Main Study):

* Definitive diagnosis of AD for at least 6 months, stringently diagnosed using the ADVN Standard Diagnostic Criteria, and has lesional skin present OR is a non-atopic healthy control subject with no personal or family history of food allergy, AD, asthma, or allergic rhinitis
* Residing in the US.

Inclusion Criteria (Sub-Study):

* Definitive diagnosis of typical plaque psoriasis for at least 6 months, stringently diagnosed using the ADVN Standard Diagnostic Criteria; or is an AD or non-atopic healthy control subject participating in the main protocol ADVN CATH 03.
* Residing in the US.

Exclusion Criteria (Main Study):

* Presence of atopy without stringent AD features, allowing only a presumptive diagnosis of AD
* Presence of AD with exfoliative erythroderma
* Presence of psoriasis
* Pregnant or lactating females
* Existence of ongoing dental disease (e.g., gingivitis)
* History of bleeding disorders
* Presence of severe AD that would be exacerbated by withholding of topical corticosteroids, oral or topical antibiotics, topical or systemic antihistamines, oral antivirals, immune enhancers (e.g., imiquimod), or topical calcineurin inhibitors within 7 days of Study Visit 2 (Baseline) and throughout the course of the trial
* Receiving systemic immunosuppressives, chemotherapeutic agents, anti-inflammatory biologics (e.g., alefacept, etanercept), systemic, oral, injectable or inhaled steroids, vitamin D supplements (more than 400 IU daily) or oral calcineurin inhibitors 30 days prior to the Study Visit 2 (Baseline) or anytime during the course of the trial
* Using topical corticosteroids, oral or topical antibiotics, oral antivirals, immune enhancers (e.g., imiquimod), topical or systemic antihistamines, or topical calcineurin inhibitors within 7 days of Study Visit 2 (Baseline) and during the course of the trial
* Receiving phototherapy (e.g., UVB, psoralen plus ultraviolet light A [PUVA]) within 30 days of Study Visit 2 (Baseline) and during the course of the trial
* Having autoimmune or immunodeficiency disease
* Presence of active systemic fungal (excluding nail fungus), bacterial, or viral infections
* History of or presence of active systemic malignancy, excluding uncomplicated non-melanoma skin cancer
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
* Inability or unwillingness of a participant to give written informed consent
* Diabetes
* Certain screening laboratory values not within normal limits, which would include calcium, serum PTH, and serum creatinine
* History of kidney disease or kidney stones
* Currently taking barbiturates such as phenobarbital (Luminal)
* Currently taking carbamazine (Tegretol), digoxin, phenytoin (Dilantin) or fosphenytoin (cerebyx)
* Currently taking diuretics such as thiazide diuretics, calcium channel blockers, or beta-blockers
* Currently taking magnesium-containing antacids, mineral oil, cholestyramine (Questran), colestipol(Colestid), orlistat (xenical), the fat substitute Olestra, cod liver oil, fish oil, or omega 3 fatty acids
* Currently taking oral antifungals such as ketoconazole
* History of serious or life-threatening anaphylactic reaction to tape or adhesives
* Lidocaine allergy
* History of or active hyperparathyroidism, sarcoid, tuberculosis or lymphoma.

Exclusion Criteria (Sub-Study):

* Presence of AD with exfoliative erythroderma
* Presence of psoriasis with exfoliative erythroderma or presence of guttate psoriasis, primary palmoplantar psoriasis, or pustular psoriasis
* Pregnant or lactating females
* Existence of ongoing dental disease (e.g., gingivitis)
* History of bleeding disorders
* Presence of psoriasis that would be severely exacerbated by withholding topical corticosteroids, oral or topical antibiotics, topical or systemic antihistamines, oral antivirals, immune enhancers (e.g.,imiquimod), or topical calcineurin inhibitors within 7 days of Study Visit 2 (Baseline) and throughout the course of the trial
* Receiving systemic immunosuppressives, chemotherapeutic agents, anti-inflammatory biologics (e.g., alefacept, etanercept), systemic, oral, injectable, or inhaled steroids, vitamin D supplements (more than 400 IU daily), or oral calcineurin inhibitors, 30 days prior to the Study Visit 2 (Baseline) or anytime during the course of the trial
* Using topical corticosteroids, oral or topical antibiotics, oral antivirals, immune enhancers (e.g., imiquimod), topical or systemic antihistamines, or topical calcineurin inhibitors within 7 days of Study Visit 2 (Baseline) and during the course of the trial
* Receiving phototherapy (e.g., UVB, psoralen plus ultraviolet light A [PUVA]) within 30 days of Study Visit 2 (Baseline) and during the course of the trial
* Having autoimmune or immunodeficiency disease
* Presence of active systemic fungal (excluding nail fungus), bacterial, or viral infections
* History of or presence of active systemic malignancy, excluding uncomplicated non-melanoma skin cancer
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
* Inability or unwillingness of a participant to give written informed consent
* Diabetes
* Screening laboratory values not within normal limits, which would include calcium, serum PTH, and serum creatinine
* History of kidney disease or kidney stones
* Currently taking barbiturates such as phenobarbital (Luminal)
* Currently taking carbamazepine (Tegretol), digoxin, phenytoin (Dilantin) or fosphenytoin (cerebyx)
* Currently taking diuretics such as thiazide diuretics, calcium channel blockers, or beta-blockers
* Currently taking magnesium-containing antacids, mineral oil, cholestyramine (Questran), colestipol (Colestid), orlistat (xenical), the fat substitute Olestra, cod liver oil, fish oil, or omega 3 fatty acids
* Currently taking oral antifungals such as ketoconazole
* History of serious or life-threatening anaphylactic reaction to tape or adhesives
* Lidocaine allergy
* History of or active hyperparathyroidism, sarcoid, tuberculosis or lymphoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gallo, MD, PhD, Study Chair — University of California, San Diego
Locations (3):
- United States (3):
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Schauber J, Dorschner RA, Yamasaki K, Brouha B, Gallo RL. Control of the innate epithelial antimicrobial response is cell-type specific and dependent on relevant microenvironmental stimuli. Immunology. 2006 Aug;118(4):509-19. doi: 10.1111/j.1365-2567.2006.02399.x. PMID 16895558
- [Result] Hata TR, Audish D, Kotol P, Coda A, Kabigting F, Miller J, Alexandrescu D, Boguniewicz M, Taylor P, Aertker L, Kesler K, Hanifin JM, Leung DY, Gallo RL. A randomized controlled double-blind investigation of the effects of vitamin D dietary supplementation in subjects with atopic dermatitis. J Eur Acad Dermatol Venereol. 2014 Jun;28(6):781-9. doi: 10.1111/jdv.12176. Epub 2013 May 3. PMID 23638978
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY14 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY14 — ImmPort study identifier is SDY14.
- Available data/document: Study Protocol: SDY14 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY14 — ImmPort study identifier is SDY14.
- Available data/document: Study summary, -design, -assessments, -adverse events, -intervention(s), -study files et al.: SDY14 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY14 — ImmPort study identifier is SDY14.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 2009 to November 2009, three centers in the United States recruited participants 18 to 70 years of age who fulfilled eligibility criteria. Refer to the Eligibility section for more details.
Groups:
- Vitamin D (Non-AD): Healthy Volunteer participants who did not have atopic dermatitis (Non-AD) and received a 21-day course of oral vitamin D3 (cholecalciferol, 4,000 international units [IU] daily).
- Vitamin D (AD): Participants classified as atopic dermatitis (AD) as defined by the Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria. Participants received a 21-day course of oral vitamin D3 (cholecalciferol, 4,000 IU daily).
- Vitamin D (Psoriasis): Participants classified as psoriasis as defined by the ADVN Standard Diagnostic Criteria. Participants received a 21-day course of oral vitamin D3 (cholecalciferol, 4,000 IU daily).
- Placebo (Non-AD): Healthy Volunteer participants who did not have AD (Non-AD) and received a 21-day course of oral vitamin D3-placebo.
- Placebo (AD): Participants classified as atopic dermatitis (AD) as defined by the Atopic Dermatitis and Vaccinia Network (ADVN) Standard Diagnostic Criteria. Participants received a 21-day course of oral vitamin D3- placebo.
- Placebo (Psoriasis): Participants classified as psoriasis as defined by the ADVN Standard Diagnostic Criteria. Participants received a 21-day course of oral vitamin D3-placebo.
Period: Overall Study
Arm/Group | Vitamin D (Non-AD) | Vitamin D (AD) | Vitamin D (Psoriasis) | Placebo (Non-AD) | Placebo (AD) | Placebo (Psoriasis)
Started | 16 | 16 | 8 | 16 | 18 | 8
Completed | 15 | 15 | 8 | 15 | 15 | 8
Not Completed | 1 | 1 | 0 | 1 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D (Non-AD) | Vitamin D (AD) | Vitamin D (Psoriasis) | Placebo (Non-AD) | Placebo (AD) | Placebo (Psoriasis) | Total
Number analyzed (Participants) | 16 | 16 | 8 | 16 | 18 | 8 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (12.3) | 32.2 (10.5) | 40.5 (11.6) | 32.2 (8.9) | 28.6 (9.8) | 37.1 (11.4) | 32.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 4 | 9 | 7 | 4 | 44
  Male | 7 | 5 | 4 | 7 | 11 | 4 | 38
Race/Ethnicity, Customized [Number; unit: Participants] — Race (Reference: Public Health Service [PHS] 398/2590, Revised 6/2009)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 4 | 1 | 1 | 2 | 2 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black | 2 | 1 | 0 | 2 | 4 | 0 | 9
    White | 12 | 9 | 6 | 11 | 11 | 5 | 54
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Other | 2 | 2 | 1 | 2 | 1 | 1 | 9
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity (Reference: Public Health Service [PHS] 398/2590, Revised 6/2009)
  Participants
    Hispanic or Latino | 4 | 1 | 1 | 2 | 0 | 1 | 9
    Not Hispanic or Latino | 12 | 15 | 7 | 14 | 18 | 7 | 73
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 8 | 16 | 18 | 8 | 82
Body Mass Index (BMI; kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — BMI is a number calculated from a person's height and weight that provides a reliable indicator of body fatness for most people. Higher values reflect greater amount of body fat. [1] In adults, a BMI less than 18.5 is underweight; 18.5 to 24.9 is a normal or healthy weight; greater than or equal to 25.0 is overweight. The height and weight was collected at baseline only.
  [1]: Healthy Weight, Assessing Your Weight, Body Mass Index http://www.cdc.gov/healthyweight/assessing/bmi/index.html
  kg/m^2 | 24.6 (5.5) | 25.2 (4.7) | 28 (6.9) | 24.5 (5.0) | 24.9 (3.5) | 27.1 (4.6) | 25.3 (4.9)
Fitzpatrick Skin Scale [Number; unit: Participants] — This scale classifies skin type categorically based on an individual's genetic disposition and skin's response to sun exposure.
  Participants
    Extremely Fair Skin | 1 | 1 | 0 | 0 | 1 | 0 | 3
    Fair Skin | 4 | 2 | 4 | 5 | 3 | 2 | 20
    Medium Skin | 4 | 5 | 2 | 4 | 7 | 4 | 26
    Olive Skin | 5 | 7 | 2 | 5 | 2 | 1 | 22
    Moderately Brown Skin | 0 | 0 | 0 | 0 | 3 | 1 | 4
    Markedly Black Skin | 2 | 1 | 0 | 2 | 1 | 0 | 6
    Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
Serum Vitamin D 25-Hydroxy (ng/mL) [Mean (Standard Deviation); unit: ng/mL] — Measurement of the amount of Vitamin D in the blood. The normal range used for our study is between 20 and 80 ng/mL.
  ng/mL | 28.8 (13.9) | 27.9 (9.7) | 31.3 (8.5) | 30.4 (11.2) | 29.3 (12.2) | 28.3 (10.7) | 29.2 (11.2)
Serum Creatinine (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Creatinine level in the blood is used as a measurement of kidney function. The normal range used for our study is 0.4 to 1.2 mg/dL.
  mg/dL | 0.8 (0.1) | 0.8 (0.1) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.1) | 0.8 (0.2)
Serum Parathyroid Hormone (pg/mL) [Mean (Standard Deviation); unit: pg/mL] — Serum Parathyroid hormone level in the blood is a measure of parathyroid gland function. The normal range used for our study is between 15 and 75 pg/mL.
  pg/mL | 37.2 (11.8) | 37.8 (13.7) | 27.6 (7.2) | 31.4 (11.8) | 34.2 (8.6) | 35.6 (12.6) | 34.4 (11.4)
Serum Calcium (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Measurement of the amount of calcium in the blood. The normal range used for our study is between 8.4 and 10.2 mg/dL.
  mg/dL | 9.3 (0.3) | 9.4 (0.4) | 9.4 (0.4) | 9.3 (0.4) | 9.5 (0.3) | 9.2 (0.3) | 9.4 (0.4)
Total Serum Immunoglobulin E (IgE) [Mean (Standard Deviation); unit: kU/L] — Total amount of IgE in the blood, which is a measurement of allergen sensitization. Higher IgE is indicative of greater allergen sensitization. There is no "normal" level for total serum IgE since a wide overlap exists between the total serum IgE in healthy non-allergic and allergic individuals.
  kU/L | 68.4 (127.3) | 1870.1 (3310.5) | 85.1 (82.0) | 45.7 (58.8) | 724.9 (2030.6) | 69.7 (109.0) | 553.3 (1825.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of CAMP mRNA in Lesional and Non-Lesional Skin for Atopic Dermatitis (AD) Participants Who Received Oral Vitamin D3 Versus Vitamin D3-Placebo
Description: Cathelicidin (CAMP) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. Cathelicidin amount is clinically significant as it is necessary to resist infection. Cathelicidin amount is not known to be clinically relevant to the clinical signs of dermatitis associated with AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (AD) | Placebo (AD)
Number analyzed (Participants) | 15 | 15
Cycle Number
  Lesional Skin Type | -0.4 (2.8) | 0.1 (2.4)
  Non-Lesional Skin Type | -0.6 (2.0) | 0.7 (2.5)
Statistical Analysis 1: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether the change in CAMP expression in lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.7, ANOVA; P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether the change in CAMP mRNA expression in non-lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.12, ANOVA; P-value is not adjusted for multiple comparisons

2. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of CAMP mRNA in Non-Lesional Skin for Non-Atopic Dermatitis (Non-AD) Participants Who Received Oral Vitamin D3 Versus Vitamin D3-Placebo
Description: Cathelicidin (CAMP) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. Non-AD is defined as a healthy volunteer without atopic dermatitis, therefore the lesional skin-type was not measured in this group. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. Cathelicidin amount is clinically significant as it is necessary to resist infection. Cathelicidin amount is not known to be clinically relevant to the clinical signs of dermatitis associated with AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Non-AD) | Placebo (Non-AD)
Number analyzed (Participants) | 15 | 15
Cycle Number | 1.2 (2.4) | 0.3 (1.7)
Statistical Analysis 1: Comparison: Vitamin D (Non-AD) vs Placebo (Non-AD); Testing whether the change in CAMP mRNA expression in non-lesional skin of Non-AD participants differs by treatment group; Test type: Superiority or Other; p = 0.3, ANOVA; P-value is not adjusted for multiple comparisons

3. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of CAMP mRNA in Lesional and Non-Lesional Skin for Psoriatic Participants Who Received Vitamin D3 Versus Vitamin D3-Placebo
Description: Cathelicidin (CAMP) messenger ribonucleic acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline, Cathelicidin abundance in psoriasis has been hypothesized to correlate with increased inflammation. No direct clinical correlation is known.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Psoriasis) | Placebo (Psoriasis)
Number analyzed (Participants) | 8 | 8
Cycle Number
  Lesional Skin Type | -0.9 (3.0) | 0.2 (3.2)
  Non-Lesional Skin Type | -0.6 (2.3) | 0.7 (2.4)
Statistical Analysis 1: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in CAMP mRNA expression in lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 0.4, ANOVA; P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in CAMP mRNA expression in non-lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 0.2, ANOVA; P-value is not adjusted for multiple comparisons

4. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of HBD-3 mRNA in Lesional and Non-Lesional Skin for Atopic Dermatitis (AD) Participants Who Received Oral Vitamin D3 Versus Vitamin D3-Placebo
Description: Human Beta-defensin 3 (HBD-3) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies as measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. HBD-3 amount is clinically significant as it is necessary to resist infection. HBD-3 amount is not known to be clinically relevant to the clinical signs of dermatitis associated with AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (AD) | Placebo (AD)
Number analyzed (Participants) | 15 | 15
Cycle Number
  Lesional Skin Type | -0.1 (7.3) | -0.8 (2.8)
  Non-Lesional Skin Type | -0.1 (3.5) | 1.4 (3.9)
Statistical Analysis 1: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether change in HBD-3 mRNA expression in lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.8, ANOVA; P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether change in HBD-3 mRNA expression in non-lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.2, ANOVA; P-value is not adjusted for multiple comparisons

5. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of HBD-3 mRNA in Non-Lesional Skin for Non-Atopic Dermatitis (Non-AD) Participants Who Received Oral Vitamin D3 Versus Vitamin D3-Placebo
Description: Human Beta-defensin 3 (HBD-3) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. Non-AD is defined as a healthy volunteer without atopic dermatitis, therefore the lesional skin-type was not measured in this group. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. HBD-3 amount is clinically significant as it is necessary to resist infection. HBD-3 amount is not known to be clinically relevant to the clinical signs of dermatitis associated with AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Non-AD) | Placebo (Non-AD)
Number analyzed (Participants) | 15 | 15
Cycle Number | 0.2 (2.8) | 1.2 (3.2)
Statistical Analysis 1: Comparison: Vitamin D (Non-AD) vs Placebo (Non-AD); Testing whether change in HBD-3 mRNA expression in non-lesional skin of Non-AD participants differs by treatment group; Test type: Superiority or Other; p = 0.4, ANOVA — P-value is not adjusted for multiple comparisons

6. Primary Outcome: Change From Baseline on Day 21 in Relative Abundance of HBD-3 mRNA in Lesional and Non-Lesional Skin for Psoriatic Participants Who Received Vitamin D3 Versus Vitamin D3-Placebo
Description: Human Beta-defensin 3 (HBD-3) Messenger Ribonucleic acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. There is no known clinical correlation between HBD-3 and psoriasis.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Psoriasis) | Placebo (Psoriasis)
Number analyzed (Participants) | 8 | 8
Cycle Number
  Lesional Skin Type | 0.8 (5.3) | -1.6 (4.4)
  Non-Lesional Skin Type | -1.5 (3.2) | -1.5 (4.3)
Statistical Analysis 1: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in HBD-3 mRNA expression in lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 0.4, ANOVA — P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in HBD-3 mRNA expression in non-lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 1.0, ANOVA — P-value is not adjusted for multiple comparisons

7. Secondary Outcome: Change From Baseline on Day 21 in Relative Abundance of IL-13 mRNA in Lesional and Non-Lesional Skin for Atopic Dermatitis (AD) Participants Who Received Vitamin D3 Versus Vitamin D3-Placebo
Description: Cytokine interleukin-13 (IL-13) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. A decrease in IL-13 may be clinically correlated with improvement of AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (AD) | Placebo (AD)
Number analyzed (Participants) | 15 | 15
Cycle Number
  Lesional Skin Type | -0.7 (2.8) | 1.1 (2.7)
  Non-Lesional Skin Type | -0.8 (2.3) | -0.1 (3.2)
Statistical Analysis 1: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether change in IL-13 mRNA expression in lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.2, ANOVA — P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (AD) vs Placebo (AD); Testing whether change in IL-13 mRNA expression in non-lesional skin of AD participants differs by treatment group; Test type: Superiority or Other; p = 0.5, ANOVA — P-value is not adjusted for multiple comparisons

8. Secondary Outcome: Change From Baseline on Day 21 in Relative Abundance of IL-13 mRNA in Non-Lesional Skin for Non-Atopic Dermatitis (Non-AD) Participants Who Received Vitamin D3 Versus Vitamin D3-Placebo
Description: Cytokine interleukin-13 ( IL-13) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. Non-AD is defined as a healthy volunteer without atopic dermatitis. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. A decrease in IL-13 may be clinically correlated with improvement of AD.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Non-AD) | Placebo (Non-AD)
Number analyzed (Participants) | 15 | 15
Cycle Number | 0.2 (2.4) | 0.5 (1.5)
Statistical Analysis 1: Comparison: Vitamin D (Non-AD) vs Placebo (Non-AD); Testing whether change in IL-13 mRNA expression in non-lesional skin of Non-AD participants differs by treatment group; Test type: Superiority or Other; p = 0.7, ANOVA — P-value is not adjusted for multiple comparisons

9. Secondary Outcome: Change From Baseline on Day 21 in Relative Abundance of IL-13 mRNA in Lesional and Non-Lesional Skin for Psoriatic Participants Who Received Vitamin D3 Versus Vitamin D3-Placebo
Description: Cytokine interleukin-13 ( IL-13) Messenger Ribonucleic Acid (mRNA) expression from skin biopsies measured by quantitative real time polymerase chain reaction (qRT-PCR). Average delta cycle threshold (CT) adjusted for non-atopic average at baseline on the arithmetic scale = [(average of (CT for CAMP - CT for Glyceraldehyde-3-phosphate dehydrogenase (GAPDH)) across replicates) - (the average of (CT for CAMP - CT for GAPDH) for non-atopic subjects at baseline)]. A negative value indicates a drop from baseline and a positive value indicates an increase from baseline. There is no known clinical correlation between IL-13 and psoriasis.
Time Frame: Baseline to Day 21
Measure: Mean (Standard Deviation); unit: Cycle Number
Arm/Group | Vitamin D (Psoriasis) | Placebo (Psoriasis)
Number analyzed (Participants) | 8 | 8
Cycle Number
  Lesional Skin Type | -2.1 (4.6) | -0.1 (4.1)
  Non-Lesional Skin Type | -0.3 (2.7) | 0.9 (3.3)
Statistical Analysis 1: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in IL-13 mRNA expression in lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 0.2, ANOVA — P-value is not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Vitamin D (Psoriasis) vs Placebo (Psoriasis); Testing whether change in IL-13 mRNA expression in non-lesional skin of psoriatic participants differs by treatment group; Test type: Superiority or Other; p = 0.3, ANOVA — P-value is not adjusted for multiple comparisons

ADVERSE EVENTS:
Description: There were no serious adverse events. No adverse events occurred at a 5% or greater frequency threshold.
Arm/Group | Vitamin D (Non-AD) | Vitamin D (AD) | Vitamin D (Psoriasis) | Placebo (Non-AD) | Placebo (AD) | Placebo (Psoriasis)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/8 | 0/16 | 0/18 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/8 | 0/16 | 0/18 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No